CLINICAL TRIAL: NCT05182632
Title: Feasibility, Acceptability and Effects of a Tele-rehabilitation Pelvic Floor Muscle Training Group Program for Urinary Incontinence in Older Women
Brief Title: Tele-rehabilitation Group Program for Urinary Incontinence in Older Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); Réseau québécois de recherche sur le vieillissement (RQRV) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER VN 20-21-33
Record Dates: First submitted 2021-09-21; First posted 2022-01-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence; Urinary Stress Incontinence
Keywords: female; aging; physiotherapy; physical therapy; pelvic floor; rehabilitation; telerehabilitation
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study
Masking Description: N/A (single-arm study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group pelvic floor tele-rehabilitation (Experimental): 12 weekly treatment online sessions + daily home exercise program
  Interventions: Behavioral: Group pelvic floor telerehabilitation

INTERVENTIONS:
Behavioral: Group pelvic floor telerehabilitation — Multimodal group physiotherapy: 12 weeks of weekly group physiotherapy treatments including education and pelvic floor muscle exercises delivered online + home exercise program

SUMMARY:
The recommended treatment for urinary incontinence (UI) in women is individualized pelvic floor muscle training (PFMT), a costly and resource-intensive approach; one Canada is currently unable to meet.

A recent non-inferiority randomized controlled trial just confirmed that group-based PFMT is equally effective but less resource-intensive (more cost-effective) than individual PFMT to treat UI in older women (ClinicalTrials.gov Identifier: NCT02039830). In times of COVID-19 however, with the Quebec, Canada's public health authorities preventing gatherings to stop the virus' spread, the potential of in-person group approaches is temporarily limited. It is thus important to develop innovative ways to deliver this first-line treatment remotely, particularly for those confined at home for whom UI can have a detrimental impact on physical health and quality of life. Ensuring an online option for group-based PFMT would also allow to increase the accessibility of UI treatment for women living in rural or remote areas in Canada, where pelvic floor rehabilitation services are not available or scarce.

To this end, this study will assess the feasibility, acceptability and effects of a tele-rehabilitation PFMT group program for UI in older women.

ELIGIBILITY:
Inclusion Criteria:

1. 65 or older, as older women will show a particular genitourinary profile compared with younger women, notably due to menopause. This age cut-off was used in other studies in UI;
2. Ambulatory (able to walk, move about safely and autonomously without any mobility device);
3. Describe a pattern of stress/mixed UI, confirmed using the Questionnaire for Incontinence Diagnosis (QUID);
4. Have at least three urinary leakage per week, persisting for 3 months or more;
5. Understand French or English instructions;
6. Report no important cognitive deficit (determined with a Mini-Mental State Evaluation (MMSE) score of 24/30 or more);
7. Have an internet access; and
8. Able to give informed consent and complete a gynecological examination and fill 7-day bladder diaries and questionnaires.

Exclusion Criteria:

1. Present risk factors known to interfere with the effects of PFMT or with the PFM evaluation, including chronic constipation (as defined by the International Working Committee for Chronic Constipation), important pelvic organ prolapse (Baden-Walker score > stage 2), or any other comorbidities with a potential impact on the treatment (i.e. cognitive impairment, diabetes, active cancer, respiratory or cardiovascular conditions, etc);
2. Currently taking medication for UI or medications affecting skeletal muscles;
3. Considered obese with a body mass index (BMI) over 35;
4. Had an active urinary or vaginal infection in the past 3 months;
5. Underwent a change in hormonal replacement therapy in the past 6 months;
6. Received pelvic floor physiotherapy treatment or surgery for UI or pelvic organ prolapse in the past year

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
number of UI episodes | at recruitment (PRE1)
  number of UI episodes, evaluated with a 7-day bladder diary
number of UI episodes | just before the intervention (PRE2)
  number of UI episodes, evaluated with a 7-day bladder diary
number of UI episodes | immediately after the 12-week intervention (POST)
  number of UI episodes, evaluated with a 7-day bladder diary
number of UI episodes | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  number of UI episodes, evaluated with a 7-day bladder diary
percentage reduction (%) in the number of UI episodes | at recruitment (PRE1), just before the intervention (PRE2), immediately after the 12-week intervention (POST), 6 months after the end of the 12-week intervention (FOLLOW-UP)
  percentage reduction (%) in the number of UI episodes, evaluated with a 7-day bladder diary

SECONDARY OUTCOMES:
urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment (PRE1)
  urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome, evaluated using the International Consultation on Incontinence Questionnaire module on UI symptoms (ICIQ-UI) short form (0-21 overall score, with higher scores indicating more sever symptoms)
urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome | just before the intervention (PRE2)
  urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome, evaluated using the International Consultation on Incontinence Questionnaire module on UI symptoms (ICIQ-UI) short form (0-21 overall score, with higher scores indicating more sever symptoms)
urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome | immediately after the 12-week intervention (POST)
  urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome, evaluated using the International Consultation on Incontinence Questionnaire module on UI symptoms (ICIQ-UI) short form (0-21 overall score, with higher scores indicating more sever symptoms)
urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome, evaluated using the International Consultation on Incontinence Questionnaire module on UI symptoms (ICIQ-UI) short form (0-21 overall score, with higher scores indicating more sever symptoms)
Changes in urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment (PRE1), just before the intervention (PRE2), immediately after the 12-week intervention (POST), 6 months after the end of the 12-week intervention (FOLLOW-UP)
  urinary symptoms and degree to which UI-associated symptoms are troubling or bothersome, evaluated using the International Consultation on Incontinence Questionnaire module on UI symptoms (ICIQ-UI) short form (0-21 overall score, with higher scores indicating more sever symptoms)
bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome | at recruitment (PRE1)
  bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome, evaluated using the Australian Pelvic Floor Questionnaire (APFQ) (0-45 score for bladder symptoms, 0-34 score for bowel symptoms, 0-15 score for pelvic organ prolapse symptoms, and 0-21 score for sexual function symptoms, with higher scores indicating more severe symptoms)
bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome | just before the intervention (PRE2)
  bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome, evaluated using the Australian Pelvic Floor Questionnaire (APFQ) (0-45 score for bladder symptoms, 0-34 score for bowel symptoms, 0-15 score for pelvic organ prolapse symptoms, and 0-21 score for sexual function symptoms, with higher scores indicating more severe symptoms)
bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome | immediately after the 12-week intervention (POST)
  bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome, evaluated using the Australian Pelvic Floor Questionnaire (APFQ) (0-45 score for bladder symptoms, 0-34 score for bowel symptoms, 0-15 score for pelvic organ prolapse symptoms, and 0-21 score for sexual function symptoms, with higher scores indicating more severe symptoms)
bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome, evaluated using the Australian Pelvic Floor Questionnaire (APFQ) (0-45 score for bladder symptoms, 0-34 score for bowel symptoms, 0-15 score for pelvic organ prolapse symptoms, and 0-21 score for sexual function symptoms, with higher scores indicating more severe symptoms)
Changes in bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome | at recruitment (PRE1), just before the intervention (PRE2), immediately after the 12-week intervention (POST), 6 months after the end of the 12-week intervention (FOLLOW-UP)
  bladder, bowel, pelvic organ prolapse and sexual function symptoms and degree to which these symptoms are troubling or bothersome, evaluated using the Australian Pelvic Floor Questionnaire (APFQ) (0-45 score for bladder symptoms, 0-34 score for bowel symptoms, 0-15 score for pelvic organ prolapse symptoms, and 0-21 score for sexual function symptoms, with higher scores indicating more severe symptoms)
UI-related quality of life | at recruitment (PRE1)
  UI-related quality of life, evaluated using the International Consultation on Incontinence Questionnaire module on Lower Urinary Tract Symptoms quality of life (ICIQ-LUTS QoL) (19-76 overall score with greater values indicating increased impact on quality of life)
UI-related quality of life | just before the intervention (PRE2)
  UI-related quality of life, evaluated using the International Consultation on Incontinence Questionnaire module on Lower Urinary Tract Symptoms quality of life (ICIQ-LUTS QoL) (19-76 overall score with greater values indicating increased impact on quality of life)
UI-related quality of life | immediately after the 12-week intervention (POST)
  UI-related quality of life, evaluated using the International Consultation on Incontinence Questionnaire module on Lower Urinary Tract Symptoms quality of life (ICIQ-LUTS QoL) (19-76 overall score with greater values indicating increased impact on quality of life)
UI-related quality of life | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  UI-related quality of life, evaluated using the International Consultation on Incontinence Questionnaire module on Lower Urinary Tract Symptoms quality of life (ICIQ-LUTS QoL) (19-76 overall score with greater values indicating increased impact on quality of life)
Changes in UI-related quality of life | at recruitment (PRE1), just before the intervention (PRE2), immediately after the 12-week intervention (POST), 6 months after the end of the 12-week intervention (FOLLOW-UP)
  UI-related quality of life, evaluated using the International Consultation on Incontinence Questionnaire module on Lower Urinary Tract Symptoms quality of life (ICIQ-LUTS QoL) (19-76 overall score with greater values indicating increased impact on quality of life)
UI-associated costs | at recruitment (PRE1)
  UI-associated costs, using the adapted Dowell-Bryant Incontinence Cost Index (DBICI) questionnaire
UI-associated costs | immediately after the 12-week intervention (POST)
  UI-associated costs, using the adapted Dowell-Bryant Incontinence Cost Index (DBICI) questionnaire
UI-associated costs | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  UI-associated costs, using the adapted Dowell-Bryant Incontinence Cost Index (DBICI) questionnaire
technology self-efficacy | at recruitment (PRE1)
  technology self-efficacy, evaluated using the Online Technologies Self-efficacy Scale (OTSES) questionnaire (30-120 overall score, with higher scores indicating lower level of technology self-efficacy)
technology self-efficacy | immediately after the 12-week intervention (POST)
  technology self-efficacy, evaluated using the Online Technologies Self-efficacy Scale (OTSES) questionnaire (30-120 overall score, with higher scores indicating lower level of technology self-efficacy)
technology self-efficacy | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  technology self-efficacy, evaluated using the Online Technologies Self-efficacy Scale (OTSES) questionnaire (30-120 overall score, with higher scores indicating lower level of technology self-efficacy)
UI related self-efficacy | at recruitment (PRE1)
  UI related self-efficacy, evaluated using the geriatric self-efficacy scale (GES) (0-120 overall score, with higher scores indicating higher level of self-efficacy related to urinary incontinence)
UI related self-efficacy | immediately after the 12-week intervention (POST)
  UI related self-efficacy, evaluated using the geriatric self-efficacy scale (GES) (0-120 overall score, with higher scores indicating higher level of self-efficacy related to urinary incontinence)
UI related self-efficacy | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  UI related self-efficacy, evaluated using the geriatric self-efficacy scale (GES) (0-120 overall score, with higher scores indicating higher level of self-efficacy related to urinary incontinence)
Pelvic floor muscles related self-efficacy | at recruitment (PRE1)
  Pelvic floor muscles related self-efficacy, evaluated using the Broome's self-efficacy scale (14 items with responses ranging 0-100 for part A and 9 items with responses ranging 0-100 for part B; an overall mean self-efficacy score is calculated, also ranging 0-100)
Pelvic floor muscles related self-efficacy | immediately after the 12-week intervention (POST)
  Pelvic floor muscles related self-efficacy, evaluated using the Broome's self-efficacy scale (14 items with responses ranging 0-100 for part A and 9 items with responses ranging 0-100 for part B; an overall mean self-efficacy score is calculated, also ranging 0-100)
Pelvic floor muscles related self-efficacy | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  Pelvic floor muscles related self-efficacy, evaluated using the Broome's self-efficacy scale (14 items with responses ranging 0-100 for part A and 9 items with responses ranging 0-100 for part B; an overall mean self-efficacy score is calculated, also ranging 0-100)
Vaginal atrophy symptoms | at recruitment (PRE1)
  Vaginal atrophy symptoms, evaluated using the Atrophy Symptom Questionnaire (ASQ) (0-15 overall score, with higher scores indicating higher severity of vaginal atrophy symptoms)
Vaginal atrophy symptoms | immediately after the 12-week intervention (POST)
  Vaginal atrophy symptoms, evaluated using the Atrophy Symptom Questionnaire (ASQ) (0-15 overall score, with higher scores indicating higher severity of vaginal atrophy symptoms)
Vaginal atrophy symptoms | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  Vaginal atrophy symptoms, evaluated using the Atrophy Symptom Questionnaire (ASQ) (0-15 overall score, with higher scores indicating higher severity of vaginal atrophy symptoms)
Patient reported improvement and satisfaction | immediately after the 12-week intervention (POST)
  Patient reported improvement and satisfaction, evaluated using the patient global impression of improvement (PGI-I) index, a single-item tool to capture perceived satisfaction with treatment: "satisfied" (does not need other treatments); "unsatisfied" (would like another treatment for UI)
Patient reported improvement and satisfaction | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  Patient reported improvement and satisfaction, evaluated using the patient global impression of improvement (PGI-I) index, a single-item tool to capture perceived satisfaction with treatment: "satisfied" (does not need other treatments); "unsatisfied" (would like another treatment for UI)
Feasibility/Acceptability (reach) | through intervention completion, for 12 weeks
  Reach aspect of feasibility/acceptability, evaluated using attendance to weekly sessions
Feasibility/Acceptability (fidelity) | through intervention completion, for 12 weeks
  Fidelity aspect of feasibility/acceptability, evaluated using the integrity of the GROUP program elements delivered by the physiotherapist during each session (checklist)
Feasibility/Acceptability (dose) | through intervention completion, for 12 weeks
  Dose aspect feasibility/acceptability, evaluated using adherence to home exercises (exercises journal)
Feasibility/Acceptability (perceived usability of the technology) | immediately after the 12-week intervention (POST)
  Perceived usability of the technology from the patients' experience as an aspect of feasibility/acceptability, evaluated using the System Usability Scale (SUS) (0-100 overall score, with higher scores indicating a higher usability)
Feasibility/Acceptability (perceived usability of the technology) | 6 months after the end of the 12-week intervention (FOLLOW-UP)
  Perceived usability of the technology from the patients' experience as an aspect of feasibility/acceptability, evaluated using the System Usability Scale (SUS) (0-100 overall score, with higher scores indicating a higher usability)
Potential challenges and satisfaction with the program from the patients' perspective | immediately after the intervention (POST)
  Potential challenges and satisfaction with the program from the patients' perspective, evaluated during focus groups or interviews using an interview guide developed from the seven dimensions of the Theoretical Framework of Acceptability (TFA), three of the five Consolidated Framework for Implementation Research (CFIR) domains and additional open-ended questions on satisfaction

OTHER OUTCOMES:
Cognitive function | at recruitment (PRE1)
  Cognitive function, evaluated using the Mini-Mental State Examination (MMSE) (0-30 overall score, with scores of 24 and over indicating a normal cognitive function)
Cognitive function | at recruitment (PRE1)
  Cognitive function, evaluated using the Montreal Cognitive Assessment (MoCA) (0-30 overall score, with scores of 26 and over indicating a normal cognitive function)
Sociodemographic characteristics | at recruitment (PRE1)
  Sociodemographic characteristics, evaluated using a home-made questionnaire recording age, weight, height, living situation, marital status, education, annual income, gynecological and medical history, medication and hormones prescriptions, smoking status, along with the Questionnaire for female Urinary Incontinence Diagnosis (QUID) to determine UI type
Signs of vaginal atrophy | at recruitment (PRE1)
  Signs of vaginal atrophy, observed during a gynecological evaluation, using the vaginal atrophy index (VAI) (6-15 overall score, with lower scores indicating more severe symptoms of vaginal atrophy)
Pelvic floor muscle function | at recruitment (PRE1)
  Gynecological evaluation of pelvic floor muscle function, using the Laycock's PERFECT score (PERFECT is an acronym with P = power of the pelvic floor muscle contraction, measured with the modified Oxford 6-point scale: 0=no contraction, 1=flicker, 2=weak, 3=moderate, 4=good, and 5=strong; E = endurance of the pelvic floor muscle contraction, measured from 0 to 10 seconds, R = repetitions, measured from 0 to 10 contractions, F = fast contractions, measured as the number of fast maximal contractions over a period of 10 seconds, E = elevation of the posterior vaginal wall during the pelvic floor muscle contraction (yes/no), C = co-contraction of the lower abdominal muscles during the pelvic floor muscle contraction (yes/no), T = timing, with the presence of synchronous involuntary contraction of pelvic floor muscles on coughing (yes/no))
Signs and severity of pelvic prolapse | at recruitment (PRE1)
  Signs and severity of pelvic prolapse, observed during a gynecological evaluation, using the Baden-Walker prolapsus score (0-4 overall score, with higher scores indicating a higher severity)

CONTACTS AND LOCATIONS:
Overall Officials: Chantale Dumoulin, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Centre de recherche de l'Institut universitaire de gériatrie de Montréal (CRIUGM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request to Prof Dumoulin for researchers whose proposed use of the data has been approved by ethics committee.
  Email: chantal.dumoulin@umontreal.ca
Supporting Information: Study Protocol, CSR
Time Frame: Available from 1 year after the publication of the main findings until five years after that publication
Access Criteria: If proposed use of the data has been approved by ethics committee

REFERENCES:
- [Background] Le Berre M, Filiatrault J, Reichetzer B, Dumoulin C. Feasibility, acceptability and effects of a group pelvic floor muscle telerehabilitation program to treat urinary incontinence in older women. Digit Health. 2022 Oct 26;8:20552076221123720. doi: 10.1177/20552076221123720. eCollection 2022 Jan-Dec. PMID 36325439
- [Background] Le Berre M, Filiatrault J, Reichetzer B, Dumoulin C. Group-Based Pelvic Floor Telerehabilitation to Treat Urinary Incontinence in Older Women: A Feasibility Study. Int J Environ Res Public Health. 2023 May 11;20(10):5791. doi: 10.3390/ijerph20105791. PMID 37239520
- [Background] Le Berre M, Filiatrault J, Reichetzer B, Kairy D, Lachance C, Dumoulin C. Online Group-based Pelvic Floor Muscle Training for Urinary Incontinence in Older Women: a Pilot Study. Int Urogynecol J. 2024 Apr;35(4):811-822. doi: 10.1007/s00192-024-05728-0. Epub 2024 Feb 5. PMID 38315227